CLINICAL TRIAL: NCT00710658
Title: A Randomized Clincial Trial to Evaluate the Effects of an Internett-based Support System for Cancer Patients on Symptom Distress, Depression, and Quality of Life.
Brief Title: Internet Support for Cancer Patients
Acronym: WebChoice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Norwegian Cancer Society (Other)
Responsible Party: Principal Investigator, Cornelia Ruland, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCS 06067/001
Record Dates: First submitted 2008-07-03; First posted 2008-07-04 (Estimated); Last update posted 2013-05-23 (Estimated); Status verified 2013-05

CONDITIONS: Cancer; Breast Cancer; Prostate Cancer
Keywords: Internet support; Tailored information; Self-management; Quality of life; Online messaging; Online discussion groups
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Patients had access to the Internet support system WebChoice that allowed them to monitor symptoms over time, and provided access to evidence-based self-management options tailored to their reported symptoms as well as to a communication area where patients could ask questions to a clinical nurse specialist in cancer care and exchange experiences with other cancer patients.
  Interventions: Behavioral: WebChoice
- 2 (No Intervention): The control group receiving usual care

INTERVENTIONS:
Behavioral: WebChoice — Patients in the experimental group had over the study period access to the Internet support system WebChoice that allowed them to monitor symptoms over time, and provided access to evidence-based self-management options tailored to their reported symptoms as well as a communication area where patients could ask questions to a clinical nurse specialist in cancer care and exchange experiences with other cancer patients.
  Patients in the control group received usual care
  Other Names: Internet support
  Arms: 1

SUMMARY:
Cancer patients often experience multiple physical, functional and psychosocial symptoms, but have limited support while being at home between treatments and during rehabilitation. WebChoice is a novel Internet support system that extends traditional health services into patients' homes. The system allows patients to monitor symptoms over time, and provides access to evidence-based self-management options tailored to their reported symptoms as well as a communication area where patients can ask questions to a clinical nurse specialist in cancer care and exchange experiences with other cancer patients.

This randomized clinical trial:

1. Tests the effects of WebChoice on primary outcomes of symptom distress, quality of life, depression and health service use, and secondary outcomes of self-efficacy, social support . We will also analyze:
2. Relationships between primary and secondary outcomes;
3. How patients' symptom distress varies over time;
4. Patients' preferences for participation in decision making about symptom management
5. How patients use WebChoice, such as frequency of use, duration, most used components;
6. How patients' experience WebChoice's usefulness and ease of use;
7. Patterns and content of patients' communication with the cancer nurse and other patients.

325 cancer patients (189 breast cancer and 136 prostate cancer patients) were recruited from throughout Norway through advertisements and invitation letters and the Norwegian Cancer Registry. Patients were randomly assigned to WebChoice or the control group that received usual care. Patients are being followed with 5 repeated measures over 12 months. Data are being collected through questionnaires, from system logs, and from interviews that were conducted in subset of experimental group patients. The primary hypothesis will be tested with Repeated Measures ANCOVA techniques. The other research questions will be answered using various inferential and descriptive techniques and through content analysis of messages and transcripts of patient interviews. This study can make a significant contribution to reduce unnecessary suffering and improve the quality of life for a large group of cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years
* Starting or currently undergoing treatment for breast or prostate cancer
* Internet access at home

Exclusion Criteria:

* Patients who had received radiation on the brain as this may have affected their abilities to reliably report their symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Symptom distress | prospective, one year, repeated measures
Quality of life | prospective, one year, repeated measures
Depression | prospective, one year, repeated measures

SECONDARY OUTCOMES:
Self-efficacy | prospective, one year, repeated measures
Social support | prospective, one year, repeated measures

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia M Ruland, PhD, Principal Investigator — Rikshospitalet-Radiumhospitalet
Locations (1):
- Rikshospitalet-Radiumhospitalet, Oslo, Norway

REFERENCES:
- [Result] Ruland CM, Andersen T, Jeneson A, Moore S, Grimsbo GH, Borosund E, Ellison MC. Effects of an internet support system to assist cancer patients in reducing symptom distress: a randomized controlled trial. Cancer Nurs. 2013 Jan-Feb;36(1):6-17. doi: 10.1097/NCC.0b013e31824d90d4. PMID 22495503
- [Result] Ruland CM, Maffei RM, Borosund E, Krahn A, Andersen T, Grimsbo GH. Evaluation of different features of an eHealth application for personalized illness management support: cancer patients' use and appraisal of usefulness. Int J Med Inform. 2013 Jul;82(7):593-603. doi: 10.1016/j.ijmedinf.2013.02.007. Epub 2013 Mar 16. PMID 23507561
- [Result] Borosund E, Cvancarova M, Ekstedt M, Moore SM, Ruland CM. How user characteristics affect use patterns in web-based illness management support for patients with breast and prostate cancer. J Med Internet Res. 2013 Mar 1;15(3):e34. doi: 10.2196/jmir.2285. PMID 23454601
- [Result] Grimsbo GH, Ruland CM, Finset A. Cancer patients' expressions of emotional cues and concerns and oncology nurses' responses, in an online patient-nurse communication service. Patient Educ Couns. 2012 Jul;88(1):36-43. doi: 10.1016/j.pec.2012.01.007. Epub 2012 Feb 11. PMID 22326865
- [Result] Grimsbo GH, Finset A, Ruland CM. Left hanging in the air: experiences of living with cancer as expressed through E-mail communications with oncology nurses. Cancer Nurs. 2011 Mar-Apr;34(2):107-16. doi: 10.1097/NCC.0b013e3181eff008. PMID 20921887
- [Result] Andersen T, Ruland CM. Cancer patients' questions and concerns expressed in an online nurse-delivered mail service: preliminary results. Stud Health Technol Inform. 2009;146:149-53. PMID 19592825
- [Result] Ruland CM, Jeneson A, Andersen T, Andersen R, Slaughter L, Bente-Schjodt-Osmo, Moore SM. Designing tailored Internet support to assist cancer patients in illness management. AMIA Annu Symp Proc. 2007 Oct 11;2007:635-9. PMID 18693913
- See also: CommuniCare tools — http://www.communicaretools.org/?lang=en-US